CLINICAL TRIAL: NCT06937034
Title: Observational Retrospective CoHort Study on Practical ExperienceS of Treatment With Foslevodopa/foScaRbidopa in Advanced Parkinson's Disease
Brief Title: Study on Practical ExperienceS of Treatment With Foslevodopa/foScaRbidopa in Advanced Parkinson's Disease
Acronym: ORCHESTRA
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H25-878
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Parkinson's Disease: Advanced Parkinson Disease Patients treated with foslevodopa/foscarbidopa.

SUMMARY:
Main objective of this study is to describe the evolution of infusion settings (base, high and low infusion rates) of foslevodopa/foscarbidopa subcutaneous infusion (LDp/CDp) at different timepoints in the treatment of advanced Parkinson's disease (aPD) as captured in ONE-CRM.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with levodopa-responsive idiopathic Parkinson's Disease prescribed on LDp/CDp CSCI in routine clinical practice who have consented to be enrolled in the AbbVie Patient Support Program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Parkinson Disease Patients treated with foslevodopa/foscarbidopa.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean Base Infusion Rate | Through end of optimization period (defined as no additional dose modification for at least 15 days since the last dose modification).
  Mean base infusion rate (ml/hour) will be assessed
Mean Low Infusion Rate | Through end of optimization period (defined as no additional dose modification for at least 15 days since the last dose modification).
  Mean low infusion rate (ml/hour) will be assessed
Mean High Infusion Rate | Through end of optimization period (defined as no additional dose modification for at least 15 days since the last dose modification).
  Mean high infusion rate (ml/hour) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- Medizinische Universitaet Graz /ID# 278569, Graz, Styria, Austria
- Medisch Spectrum Twente /ID# 276695, Enschede, Overijssel, Netherlands
- Universitatea De Medicină Și Farmacie Victor Babeș /ID# 276720, Timișoara, Timiș County, Romania
- Karolinska University Hospital Solna /ID# 277116, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H25-878